CLINICAL TRIAL: NCT02991638
Title: Efficacy and Safety of Ibrutinib in Patients With Chronic Lymphocytic Leukemia and Other Indolent B-cell Lymphomas Who Are Chronic Hepatitis B Virus Carriers or Occult Hepatitis B Virus Carriers
Brief Title: Efficacy and Safety of Ibrutinib in Patients With CLL and Other Indolent B-cell Lymphomas Who Are Chronic Hepatitis B Virus Carriers or Occult Hepatitis B Virus Carriers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKUBTK01
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Chronic Lymphocytic Leukemia; Indolent B-cell Lymphomas; Chronic Hepatitis B; Lymphoma, Small Lymphocytic; Mantle-Cell Lymphoma; Waldenstrom's Macroglobulinaemia; Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hepatitis B, Chronic; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Follicular | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib (Other): Relapsed / refractory chronic lymphocytic leukemia and Waldenstrom macroglobulinaemia (lymphoplasmacytic lymphoma): 420 mg daily Relapsed / refractory mantle cell lymphoma: 560 mg daily Relapsed / refractory indolent B-cell non-Hodgkin lymphoma: 560 mg daily Treatment is continued until disease progression
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Relapsed / refractory chronic lymphocytic leukemia and Waldenstrom macroglobulinaemia (lymphoplasmacytic lymphoma): 420 mg daily Relapsed / refractory mantle cell lymphoma: 560 mg daily Relapsed / refractory indolent B-cell non-Hodgkin lymphoma: 560 mg daily Treatment is continued until disease progression
  Other Names: Imbruvica

SUMMARY:
Efficacy and Safety of ibrutinib in patients with chronic lymphocytic leukemia and other indolent B-cell lymphomas who are chronic hepatitis B virus carriers or occult hepatitis B virus carriers

DETAILED DESCRIPTION:
Ibrutinib is a selective oral Burton tyrosine kinase inhibitor. Through interfering with the downstream pathways of B-cell receptor signaling, it inhibits proliferation and induces apoptosis in many B-cell lymphoid malignancies. The clinical benefit of ibrutinib has been demonstrated in patients with relapsed/refractory chronic lymphocytic leukaemia, mantle cell lymphoma, small lymphocytic lymphoma, and other indolent B-cell non-Hodgkin lymphomas.

The pivotal trials of ibrutinib excluded HBsAg+ patients. Therefore, the effects of ibrutinib on HBsAg+ and anti-HBc+ patients remain entirely undefined. In view of the B-cell signaling inhibitory activity of ibrutinib, which might be more potent than rituximab in suppressing B-cells, HBV reactivation in patients exposed previously to HBV infection, including chronic HBV carriers and occult HBV carriers, could be a major clinical problem.

To enable ibrutinib to be prescribed in Asia and other regions of the world where HBV is endemic, evidence-based recommendations on prevention of HBV reactivation in at-risk populations, including chronic HBV carriers (HBsAg+), and occult HBV carriers (HBsAg- but anti-HBc+), are urgently needed.

The following treatment regimens will be adopted. Relapsed / refractory chronic lymphocytic leukemia and Waldenstrom macroglobulinaemia (lymphoplasmacytic lymphoma): 420 mg daily.

Relapsed / refractory mantle cell lymphoma: 560 mg daily. Relapsed / refractory indolent B-cell non-Hodgkin lymphoma: 560 mg daily. Treatment is continued until disease progression.

A total of 62 patients will be recruited, including 16 HBsAg+ patients, and 46 occult HBV carriers

Sample size calculation of occult HBV carriers For occult HBV carriers, the sample size is calculated according to the following information, based on our previous observations (as detailed in reference 3). The HBV reactivation rate in HBsAg-, anti-HBc+, anti-HBs+ patients is hypothesized to be 34%, which may increase to 68% in HBsAg-, anti-HBc+, but anti-HBs- patients [3]. Assuming a power of 80% and an alpha-risk of 0.1, together with the ratio of anti-HBs+ : anti-HBs- patients to be 2:1, we expect to recruit 42 HBsAg-, anti-HBc+ patients. With a dropout rate of 10%, the total number of patients to be recruited in this group will be 46.

Sample size calculation of HBsAg+ patients For HBsAg+ patients, the sample size is calculated according to the following information, based on our previous observations (as detailed in reference 3). The ratio of occult carriers (HBsAg-, anti-HBc+) : HBsAg+ patients is about 3: 1.3 Hence, the total number of HBsAg+ to be recruited will be 14 (42 divided by 3). With a drop-out rate of 10%, the total number of patients to be recruited in this group will be 16.

Approximate breakdown of number of patients in each category to be recruited Based on our previous observations on the proportions of low-grade B-cell lymphoid malignancies,8 an approximate breakdown of number of patients is as follows: follicular lymphoma (N=32), chronic lymphocytic leukemia/small lymphocytic lymphoma (N=11), marginal zone B-cell lymphoma (N=11), mantle cell lymphoma (N=5), and Waldenstrom macroglobulinemia (N=5).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between age of 18 - 80 years
2. Patients with indolent B-cell lymphoproliferative neoplasms that have relapsed or are refractory after at least one standard line of therapy that contains rituximab
3. Pathologically proven B-cell lymphoproliferative neoplasms including chronic lymphocytic leukaemia/small lymphocytic lymphoma, mantle cell lymphoma, marginal-zone B-cell lymphoma, and Waldenstrom macroglobulinaemia (lymphoplasmacytic lymphoma).
4. Pathologically proven follicular lymphoma, with relapse or disease progression > 12 months after previous rituximab therapy.
5. Chronic HBV carriers (HBsAg+)
6. Occult HBV carriers (HBsAg-, anti-HBc+ and HBV DNA-)
7. Haematology values within the following limits:

   1. Absolute neutrophil count (ANC)1000/mm3 independent of growth factor support
   2. Platelets 100,000/mm3, or 50,000/mm3 if bone marrow is involved, and independent of transfusion support in either situation
8. Biochemical values within the following limits:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 x upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
   3. Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockcroft Gault) ≥ 40 mL/min/1.73m2
9. Competent to give an informed consent

Exclusion Criteria:

1. Concomitant chronic liver diseases not related to HBV
2. Known history of drug-induced liver injury, chronic active hepatitis C infection, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, on-going extra-hepatic obstruction caused by cholelithiasis, cirrhosis of the liver and portal hypertension
3. Known history of drug induced pneumonitis
4. Known history of inflammatory bowel disease
5. Woman who are pregnant or breast-feeding
6. Patients who do not consent to the use of effective contraception during the study
7. Active infections.
8. Evidence of ongoing active HBV hepatitis (ALT and/or AST > 2x upper limit of normal, and detectable HBV DNA)
9. Patients known to have histological transformation of CLL to an aggressive lymphoma
10. Vaccinated with live, attenuated vaccines within 4 weeks of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 2 years
  proportion of patients achieving CR or partial remission (PR)
Duration of remission | two year
Rates of HBV Reactivation while on Ibrutinib therapy | two year
Adverse events and severe adverse events | two year
  Incidence of AE and SAE by severity grading as assessed according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yok Lam Kwong, MD(HK),, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided